CLINICAL TRIAL: NCT05325892
Title: Prospective Analysis of Influencing Factors of Hypotension in Diabetic Patients Undergoing Dialysis
Brief Title: Analysis of Influencing Factors of Hypotension in Diabetic Patients Undergoing Dialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200202
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Hemodialysis; Diabetes
Keywords: Intradialytic hypotension
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IDH: Diabetic patients with maintenance hemodialysis who developed hypotension during hemodialysis therapy.Intradialytic hypotension (IDH) is defined as a decrease in systolic blood pressure by ≥20 mm Hg or a decrease in MAP by ≥10 mm Hg associated with symptoms that include: abdominal discomfort; yawning; sighing; nausea; vomiting; muscle cramps; restlessness; dizziness or fainting; and anxiety.
  Interventions: Combination Product: This is an observational study
- non-IDH: Diabetic patients with maintenance hemodialysis who did not develop hypotension during hemodialysis treatment.Intradialytic hypotension (IDH) is defined as a decrease in systolic blood pressure by ≥20 mm Hg or a decrease in MAP by ≥10 mm Hg associated with symptoms that include: abdominal discomfort; yawning; sighing; nausea; vomiting; muscle cramps; restlessness; dizziness or fainting; and anxiety.
  Interventions: Combination Product: This is an observational study

INTERVENTIONS:
Combination Product: This is an observational study — This is an observational study

SUMMARY:
Hypotension (IDH) during dialysis is a common complication in hemodialysis, and the incidence is 20-50% in hemodialysis patients, the proportion of diabetic patients with IDH is 26.7%, which is much higher than that of non-diabetic patients. Currently, there are few studies on the influencing factors and related thresholds of IDH in diabetic patients.A total of 180 eligible patients were selected from Beijing Friendship Hospital, Beijing Nuclear Industry Hospital, Beijing Daxing District People's Hospital, Beijing Zhongneng Jian Hospital. General data of patients were collected. Dialysis prescription Blood pressure biochemical parameters and cardiac color ultrasound parameters were divided into IDH group and non-IDH group according to the incidence of IDH during dialysis Logistic regression was used to analyze the influencing factors of IDH, and ROC curve was used to explore the threshold of related factors.

DETAILED DESCRIPTION:
research background：According to the executive summary of 2015 annual data report of China Kidney Disease Network (CK-NET), hemodialysis is the main way of renal replacement therapy, accounting for 91.0% of all dialysis patients, and the prevalence rate of diabetic dialysis patients accounts for 26.7 of hemodialysis patients.Intradialytic hypotension (IDH) is a common complication in hemodialysis, which is related to high morbidity and mortality.There are significant differences in the incidence of IDH in patients with different diagnostic criteria, and there are also significant differences in the incidence of IDH in different populations with similar definitions.At present, Kidney Disease: Improving Global Outcomes (KDIGO) has not provided the diagnostic criteria for IDH.China's nephrology community has not reached a consensus on this.The diagnostic criteria for IDH recommended by KDOQI and European Best Practice Guidelines (EBPG) are a 20 mmHg decrease in arterial systolic blood pressure (SBP) during dialysis, or a 10 mmHg decrease in mean arterial blood pressure MmHg, accompanied by headache, malaise, convulsions, nausea, vomiting, irritability and other hypotension-related symptoms or related intervention measures during dialysis.In previous retrospective studies, it is not easy for researchers to obtain the clinical symptoms and related management measures of PATIENTS with IDH. Most retrospective studies take the value of patients' blood pressure drop as the reference standard for the occurrence of IDH, and further prospective studies are needed on the influencing factors of IDH.The majority of diabetic patients with autonomic nervous dysfunction and decreased vascular regulation are at high risk of IDH.A large number of studies have proved that IDH is more likely to occur in patients with diabetes, but there are few prospective studies on the risk factors of IDH in patients with diabetes.

By collecting the general information of diabetes patients, age of dialysis, history of coronary heart disease, history of hypertension, current antihypertensive drugs, postural hypotension, dry weight, ultrafiltration volume, ultrafiltration rate, pre-dialysis blood pressure, blood pressure during dialysis, and blood pressure after dialysis, In dialysis hypotension associated symptoms and treatment measures, albumin, hemoglobin, blood lipid, BNP, before and after dialysis, blood sugar, blood biochemical indexes such as calcium, heart colour to exceed the main parameters (EF %, E/A, aortic root diameter), statistical analysis, to explore the influence factors of hypotension in dialysis patients with diabetes and related threshold. The above examinations are all tests in the normal clinical treatment process, and the frequency and items of patients' tests will not be increased.

4. Research scheme research design prospective cohort study Research object Study population: Maintenance hemodialysis patients treated in Beijing Zhongnengjian Hospital, Beijing Daxing District People's Hospital, Beijing Friendship Hospital, Capital Medical University, From March 1, 2021 to September 30, 2022 Planned enrollment: 180 patients, including 60 patients from Beijing Friendship Hospital affiliated to Capital Medical University, 40 patients from Beijing Zhongnengjian Hospital and 40 patients from Beijing Daxing District People's Hospital Inclusion criteria: ① Diagnosis of end-stage renal disease; ② Maintenance hemodialysis >3 months; ③ Age >18; ④ Dialysis 3 times a week; ⑤ Diagnosed with diabetes Exclusion criteria: 1.① Acute renal failure; ② Acute heart failure; ③ Dialysis with ultrafiltration curve or sodium curve mode; ④ The upper limb blood pressure can not be measured ⑤ the systolic blood pressure before penetration <90mmHg; ⑥ Malignant tumor fluid state.

research process A total of 180 patients eligible for inclusion were screened from Beijing Friendship Hospital, Beijing Nuclear Industry Hospital, Beijing Daxing District People's Hospital, Beijing Zhongnengjian Hospital, Capital Medical University, and their general data from 2022-3-1 to 2022-9-30 were collected The main parameters of cardiac color ultrasound were divided into IDH group and non-IDH group according to the occurrence of IDH in dialysis. The influencing factors of IDH were analyzed by logistic regression, and the threshold of related factors of IDH was explored by ROC curve.

Observation indexes: prospective collection history of dialysis age age and gender in patients with coronary heart disease History of high blood pressure Present use of antihypertensive drugs without orthostatic hypotension dry weight, ultrafiltration volume of the ultrafiltration rate through blood pressure before dialysis after dialysis, blood pressure and blood pressure in the dialysis hypotension related symptoms and treatment measures Hemoglobin before and after the blood lipid albumin dialysis blood sugar Blood calcium, BNP and other biochemical indicators Main parameters of cardiac color ultrasound (EF% E/A aortic root diameter).

Determination of sample size: Combined with previous studies, estimate according to sample size formula.

Informed consent This study was an observational study, in which data were recorded during the diagnosis and treatment of patients, consent was solicited and informed consent was signed.

Statistical methods: SPSS20.0 statistical software was used for statistical analysis, normality test was performed for continuous variables, mean standard deviation was used for numerical variables conforming to normal distribution, T test was used for inter-group comparison, counting data was expressed as %, chi-square test was used for comparison and multivariate Logistic regression was used to analyze the gender and age of patients in the two groups Blood ALB blood Hb BNP blood lipid cardiac color ultrasound EF% E/A Blood pressure UFR dry weight in the aortic root before transportion. ROC curve was used to analyze the threshold of important factors influencing the incidence of hypotension during dialysis. 0.05 was considered statistically significant.

Quality control: This study is a prospective study. According to literature and clinical experience, patient data are collected and input into the database. Experienced doctors check and give feedback when problems are found. Develop daily plans and consistency check procedures in advance to ensure accurate, complete and comprehensive data; Identify and address errors and omissions; Keep records of relevant documents, especially the original database, to trace back the quality control activities.

ELIGIBILITY:
Inclusion Criteria:

* ① Diagnosis of end-stage renal disease; ② Maintenance hemodialysis >3 months; ③ Age >18; ④ Dialysis 3 times a week; ⑤ Diagnosed with diabetes

Exclusion Criteria:

* ① Acute renal failure; ② Acute heart failure; ③ Dialysis with ultrafiltration curve or sodium curve mode; ④ The upper limb blood pressure can not be measured ⑤ the systolic blood pressure before penetration <90mmHg; ⑥ Malignant tumor fluid state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients with maintenance hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
IDH | during dialysis
  20 mmHg decrease in arterial systolic blood pressure (SBP) during dialysis, or a 10 mmHg decrease in mean arterial blood pressure MmHg, accompanied by headache, malaise, convulsions, nausea, vomiting, irritability and other hypotension-related symptoms or related intervention measures during dialysis

CONTACTS AND LOCATIONS:
Overall Officials: zongli diao, doctor, Study Director — Beijing Friendship Hospital; peiyi zhou, doctor, Study Director — People's Hospital of Beijing Daxing District; guo liu, bachelor, Study Director — Beijing Zhongnengjian Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No